CLINICAL TRIAL: NCT04716335
Title: Neurodynamics of Prosocial Emotional Processing Following Serotonergic Stimulation With N,N-Dimethyltryptamine (DMT) and Harmine in Healthy Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Psychiatric University Hospital, Zurich (Other)
Collaborators: University of Basel (Other)
Responsible Party: Principal Investigator, Milan Scheidegger, Principal Investigator, Psychiatric University Hospital, Zurich
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2018-01385
Record Dates: First submitted 2020-12-23; First posted 2021-01-20 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Emotions; Mood; Cognitive Function 1, Social; Empathy
MeSH Terms: interventions — Harmine; N,N-Dimethyltryptamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Harmine + DMT (Experimental)
  Interventions: Drug: DMT; Drug: Harmine
- Harmine + Placebo(DMT) (Experimental)
  Interventions: Drug: Harmine; Drug: Placebo (DMT)
- Placebo(Harmin & Placebo) (Placebo Comparator)
  Interventions: Drug: Placebo (Harmine); Drug: Placebo (DMT)

INTERVENTIONS:
Drug: DMT — DMT
  Arms: Harmine + DMT
Drug: Harmine — Harmine
  Arms: Harmine + DMT; Harmine + Placebo(DMT)
Drug: Placebo (Harmine) — Placebo for Harmine
  Arms: Placebo(Harmin & Placebo)
Drug: Placebo (DMT) — Placebo for DMT
  Arms: Harmine + Placebo(DMT); Placebo(Harmin & Placebo)

SUMMARY:
The aim of the project is to assess brain network dynamics, self-referential information processing and prosociality and learning following the modulation of the serotonin-system by serotonergic-psychoactive compounds.

ELIGIBILITY:
Inclusion Criteria:

* Willing and capable to give informed consent for the participation in the study after it has been thoroughly explained
* Little or no previous experiences with psychedelic substances
* Body mass index (BMI) between 18.5 and 25
* Willing to refrain from drinking caffeine 3 days and alcohol the day before testing session, from drinking alcohol and caffeinated drinks at the testing days and from consuming psychoactive substances or other medications for 2 weeks before testing days and for the duration of the study
* Able and willing to comply with all study requirements
* Informed consent form was signed
* Good knowledge of the German language

Exclusion Criteria:

* Previous significant adverse response to a hallucinogenic drug
* Participation in another study where pharmaceutical compounds will be given
* Self or first-degree relatives with present or antecedent psychiatric disorders
* History of head trauma or fainting
* Recent cardiac or brain surgery
* Current use of medication or psychotropic substances (including nicotine addiction)
* Presence of major internal or neurological disorders (including sepsis, pheochromocytoma, thyrotoxicosis, drug-induced fibrosis, familiar or basilar artery migraine)
* Cardiovascular disease (hypertonia, coronary artery disease, heart insufficiency, myocardial infarction, coronary spastic angina)
* Peripheral vascular disease (thromboangiitis obliterans, luetic arteritis, severe arteriosclerosis, thrombophlebitis, Raynaud's disease)
* Liver or renal disease

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Change in Behavioral Outcome Measures (Social Value Orientation - SVO, Charity Donation Frank Task) | Acute drug effects (240 minutes - Charity Donation Frank Task, 300 minutes - SVO)
  Social Cognition
Change in Behavioral Outcome Measures (Visuall Oddball, Karaoke Task) | Acute drug effects (60 min - Visuall Oddball, 150 min - Karaoke Task)
  Self-referential Processing
Change in Pharmacological-EEG (Lagged Phase Synchronicity) | Baseline, Acute drug effects (30 minutes , 135 minutes, 195 minutes, 285 minutes)
  Functional brain connectivity
Change in Pharmacological-EEG (Resting State) | Baseline, Acute drug effects (30 minutes , 135 minutes, 195 minutes, 285 minutes)
  Spectral Density
Change in Pharmacological-EEG | Acute drug effects (60 minutes, 240 minutes)
  Event-Related Potentials (ERP)

SECONDARY OUTCOMES:
Change in biomarkers | Baseline, Acute drug effects (0 minutes, 30 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes, 210 minutes, 240 minutes, 270 minutes, 300 minutes)
  Tryptophan catabolites (TRYCAT)
Change in biomarkers | Baseline, Acute drug effects (30 minutes, 90 minutes, 150 minutes, 300 minutes)
  Brain-derived Neurotrophic Factor (BDNF)
Change in biomarkers | Baseline, Acute drug effects (0 minutes, 30 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes, 210 minutes, 240 minutes, 270 minutes, 300 minutes)
  Hypothalamic-Pituitary-Adrenal Axis (HPA-A)
Change in biomarkers | Baseline, Acute drug effects (0 minutes, 30 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes, 210 minutes, 240 minutes, 270 minutes, 300 minutes)
  API (DMT, Harmine)
Change in biomarkers | Baseline, Acute drug effects (30 minutes, 90 minutes, 150 minutes, 300 minutes)
  Neuroinflammation - Interleukines
Change in biomarkers | Baseline, Acute drug effects (30 minutes, 90 minutes, 150 minutes, 300 minutes)
  Oxidative Stress Markers (Nitric Oxide Synthase)
Psychometry | Baseline, Acute, 1 day after, 1 week after, 1 month after and 4 month after intervention
  Cognitive Flexibility
Psychometry | Baseline, Acute, 1 day after, 1 week after, 1 month after and 4 month after intervention
  MINDSENS
Psychometry | Baseline, Acute, 1 day after, 1 week after, 1 month after and 4 month after intervention
  PANAS
Psychometry | Baseline, Acute, 1 day after, 1 week after, 1 month after and 4 month after intervention
  CFI
Psychometry | Baseline, Acute, 1 day after, 1 week after, 1 month after and 4 month after intervention
  SRQ
Psychometry | Baseline, Acute, 1 day after, 1 week after, 1 month after and 4 month after intervention
  MBQ

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatric University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mueller MJ, Aicher HD, Dornbierer DA, Marten L, Suay D, Meling D, Elsner C, Wicki IA, Muller J, Poetzsch SN, Caflisch L, Hempe A, Steinhart CP, Puchkov M, Kost J, Landolt HP, Seifritz E, Quednow BB, Scheidegger M. Pharmacokinetics and pharmacodynamics of an innovative psychedelic N,N-dimethyltryptamine/harmine formulation in healthy participants: a randomized controlled trial. Int J Neuropsychopharmacol. 2024 Dec 28;28(1):pyaf001. doi: 10.1093/ijnp/pyaf001. PMID 39774840
- [Derived] Dornbierer DA, Marten L, Mueller J, Aicher HD, Mueller MJ, Boxler M, Kometer M, Kosanic D, von Rotz R, Puchkov M, Kraemer T, Landolt HP, Seifritz E, Scheidegger M. Overcoming the clinical challenges of traditional ayahuasca: a first-in-human trial exploring novel routes of administration of N,N-Dimethyltryptamine and harmine. Front Pharmacol. 2023 Nov 27;14:1246892. doi: 10.3389/fphar.2023.1246892. eCollection 2023. PMID 38089057